CLINICAL TRIAL: NCT02718534
Title: Effectiveness and Safeness of Early Limb Rehabilitation Therapy Within 48 h of Acute Stroke Onset: a Randomized Controlled Trial
Brief Title: Early Limb Rehabilitation Therapy Within 48 h of Acute Stroke Onset(ERTAS)
Acronym: ERTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Hongyu Zhao, deputy director of emergency department, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERTAS; LNCCC-D12-2015 (Other Grant/Funding Number: Health and family planning commission of Liaoning Province. China.)
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Time of First Rehabilitation Therapy
MeSH Terms: interventions — Stroke Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERTAS-1 (Experimental): first limb rehabilitation therapy took place within 48h for patients with acute stroke (modified Rankin Scale Score 3-4)
  Interventions: Behavioral: stroke rehabilitation
- ERTAS-2 (Active Comparator): first limb rehabilitation therapy took place after 48h for patients with acute stroke (modified Rankin Scale Score 3-4)
  Interventions: Behavioral: stroke rehabilitation

INTERVENTIONS:
Behavioral: stroke rehabilitation — Physical rehabilitation exercise between 24 and 48 hours and after 48 hours

SUMMARY:
This study aimed to evaluate effectiveness of initial limb rehabilitation compare therapy took place within 48h with therapy took place after 48h for patients with stroke (modified Rankin Scale Score 3-4).

DETAILED DESCRIPTION:
Early rehabilitation after stroke is thought to contribute to the effects of stroke-unit care. However, time of initial rehabilitation therapy is poorly defined and not underpinned by strong evidence in patients with stroke (modified Rankin Scale Score 3-4). The investigators do this parallel-group, single-blind, randomized controlled trial in shengjing hospital of China Medical University. Participants (aged≥18 years) with ischaemic or haemorrhagic stroke, first or recurrent, who meet physiological criteria are randomly assigned (1:1), to receive usual stroke therapy. Treatment with recombinant tissue plasminogen activator is allowed. Randomisation is stratified by study site and stroke severity. The primary outcome was a outcome 3 months after stroke, defined as a modified Rankin Scale score of 3-4. The investigators do analysis on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed acute stroke within 24h onset. Head CT or MRI scans were confirmed the diagnosed.
2. The age was from 18 to 75 years old.
3. Temperature ≤38.0℃，Pulse rate 60-100bpm，Respiratory rate≤24 bpm，systolic blood pressure≤220mmHg.
4. Glasgow score: 9-14.
5. Acute Physiology and Chronic Health Evaluation(APACHE Ⅱ)score: ≤17.
6. National Institutes of Health Stroke Scale (NIHSS)score: <16. (Upper and lower extremity motor function item score<8).
7. Modified Rankin Scale score:3-4.
8. There were no serious diseases before, such as heart, liver, kidney and lung diseases.
9. Patients themselves or their nominated representative sign the informed consent form.

Exclusion Criteria:

1. There were unstable vital sign. There were serious organic dysfunction (heart, liver, kidney or lung).
2. Patients with transient ischemic attack.
3. Patients with subarachnoid haemorrhage.
4. Patients with haemorrhage were documented immediate surgery.
5. Pregnancy patients with stroke.
6. During the course of the project, major diseases took place (such as, myocardial infarction, gastrointestinal bleeding, respiratory failure, pulmonary embolism, deep vein thrombosis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome was a favourable outcome at 3 months after stroke, measured with the Fugl-Meyer motor function score. | 90 days
  Fugl-Meyer score

SECONDARY OUTCOMES:
The primary outcome was a favourable outcome at 3 months after stroke, measured with Modified Rankin Scale score. | 90 days
  Modified Rankin Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhao, doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Background] AVERT Trial Collaboration group. Efficacy and safety of very early mobilisation within 24 h of stroke onset (AVERT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):46-55. doi: 10.1016/S0140-6736(15)60690-0. Epub 2015 Apr 16. PMID 25892679
- [Derived] Wang F, Zhang S, Zhou F, Zhao M, Zhao H. Early physical rehabilitation therapy between 24 and 48 h following acute ischemic stroke onset: a randomized controlled trial. Disabil Rehabil. 2022 Jul;44(15):3967-3972. doi: 10.1080/09638288.2021.1897168. Epub 2021 Mar 18. PMID 33736542